CLINICAL TRIAL: NCT01146002
Title: Language-based Learning Skills and ADHD: Impact of Treatment With Sustained-release Guanfacine
Brief Title: Language-based Learning Skills and Attention Deficit Hyperactivity Disorder (ADHD): Impact of Treatment With Sustained-release Guanfacine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurology Group of Bergen County, P.A. (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Guanfacine learning study
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder, primarily inattentive or combined type.
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guanfacine treated. (Other): Single arm - all patients treated with study drug. Comparison is against pre-treatment performance.
  Interventions: Drug: Guanfacine (sustained release)

INTERVENTIONS:
Drug: Guanfacine (sustained release) — Treated with study drug once screening and initial testing is completed (see protocol above)

SUMMARY:
This study is investigating the effect of sustained-release guanfacine (Intuniv) on language-based learning skills in children age 6-12 who are diagnosed with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
LANGUAGE-BASED LEARNING SKILLS AND ADHD: IMPACT OF TREATMENT WITH SUSTAINED-RELEASE GUANFACINE

Background:

Children with attention-deficit/hyperactivity disorder (ADHD) often do poorly in school (1,2,3). Their slow academic progress is typically attributable to inattention, restlessness, disorganization and distractibility, all of which diminish their ability to learn. Additionally, these manifestations of ADHD may worsen an underlying specific learning disability (SLD), which is a common comorbidity of ADHD (1,4,5).

Treatment for ADHD is often initiated with the goal of enhancing learning and fostering academic success. Yet changes in academic achievement resulting from the pharmacological treatment of ADHD have been less evaluated in clinical research than changes in specifically defined behaviors. Such behaviors typically include lack of attention to task, fidgeting, calling out, disorganization and hyperactivity. These behaviors, rather than overall academic improvement, are also what are measured with typical ADHD rating scales (6).

A relatively small number of clinical studies have assessed the impact of medications for the treatment of ADHD on academic progress during childhood or adolescence. Some of these studies (3,7) have focused on long-term measures, such as lack of grade retention and ultimate graduation from high school. Other research has tried to directly measure the effect of medication for ADHD on the ability to perform particular academic tasks. Typically, the ability to efficiently and correctly solve a series of arithmetical problems - first, with no treatment, and then while taking stimulant medication, has been measured (8,9). These studies have demonstrated that both methylphenidate-based and amphetamine-based stimulant drugs enable greater speed, efficiency and accuracy.

Studying arithmetical speed and accuracy to determine a medication's helpfulness in the school setting may be insufficient, however, since mathematics is not relevant to most of the academic material and skills that children are required to learn. To the investigator's knowledge no prior studies have evaluated the impact of medications for ADHD on language-based tasks such as reading or reading comprehension. Yet competency in reading, reading comprehension, auditory comprehension and writing is arguably more important than competency in arithmetic during grammar school, and becomes even more essential during middle school and high school. Moreover, even in apparently "arithmetical" subjects such as mathematics and science, word problems are often utilized, so that arithmetical ability alone is insufficient. Finally, it should also be noted that the most common forms of SLD are language-based disabilities that manifest as a weakness in reading, comprehension, or writing skill, but not arithmetical skill (10). For all these reasons, we should not assume that testing arithmetical performance is adequate to demonstrate the effectiveness of medication for ADHD, whether or not a coexisting SLD is present.

Study Protocol

This will be a single-arm study in which the language-based academic skills of children diagnosed with ADHD will be assessed prior to, and then during treatment with sustained-release guanfacine (GXR). Children will be diagnosed with ADHD using standard rating instruments (see below). Children meeting inclusion and exclusion criteria will undergo testing of language-based academic skills with the Woodcock-Johnson III test prior initiating treatment with GXR. The daily dose of GXR will then be initiated at 1 mg and titrated by 1 mg in weekly intervals, based on significant improvement in ADHD rating scales, the to a maximum dose of 4 mg. Once significant improvement in ADHD manifestations is recorded using rating scales, upward titration will stop and the dose will be maintained. After five weeks repeat testing using the WJIII will be done. Results of pre- and post-medication testing will be compared for the group using appropriate statistical methods.

Study Population:

We will attempt to recruit 20 or more children with ADHD in the setting of a well-established suburban pediatric neurology office practice.

Primary efficacy endpoint:

Statistically significant (p<0.05 level) improvement in Woodcock-Johnson test scores during treatment with GXR compared to pre-treatment.

Inclusion and exclusion criteria:

Children between the ages of 6 to 12 years with newly diagnosed ADHD-inattentive type or ADHD-combined type will be identified. The diagnosis of ADHD will be established using the Diagnostic and Statistical Manual of Mental and Related Disorder, version IV, Text Revision (DSM-IV TR, 2000) criteria and the ADHD Rating Scale IV (ADHD-RS; DuPaul et al., 1998).

Patients with any of the following are excluded:

* Intelligence (IQ) below 85 as determined by formal testing (see below).
* Identified or suspected genetic syndromes.
* Autism or other pervasive developmental disorders.
* Psychiatric disorders other than ADHD and oppositional defiant disorder.
* Heart, liver or renal disease.
* Cancer.
* Epilepsy or non-febrile seizure history.
* Cardiac arrhythmia, bradycardia, or syncope.
* Any other condition considered to be potentially exacerbated or endangered by treatment with an alpha-2 agonist drug.

  * Prior treatment with medication for ADHD will not be an exclusion criterion.

Screening and initiation of study:

Children between the ages of 6 to 12 years with newly diagnosed ADHD-inattentive type or -combined type will be identified. The diagnosis of ADHD will be made by means of the DSM-IV -TR criteria and the ADHD-RS.

Appropriate informed consent to participate in the study will be obtained from the child's parent(s).

Patients will be screened for medical conditions excluding them from the study. Vital signs will be checked; patients with values below the 2nd and above the 98th percentile will be also excluded. A comprehensive physical examination will be performed. Intelligence testing using the Wechsler Intelligence Scale for Children, 4th ed. (WISC; Wechsler, 2003) will be performed. Children with a full-scale IQ below 85 will be excluded.

There will then be a one-week period which will serve as a washout for any currently taken medication for ADHD.

Treatment with medication and testing of learning parameters:

Children qualifying for the study will be administered selected portions of the Woodcock-Johnson Test III (WJ-III; Woodcock et al., 2006). We will utilize sections of this test evaluating phonetics, reading fluency, reading comprehension and listening comprehension. Writing ability will not be assessed because of the confounding influence of fine motor development on writing speed. Mathematical ability will also not be tested.

This test includes an "A" and a "B" form. Only the A form will be used initially so as to minimize practice effect when the test is later repeated.

Treatment with GXR will be initiated immediately after testing, and titrated over a 5-week period. The initial dosage will be 1 mg daily and will be titrated in weekly intervals to a maximum dose of 4 mg. Clinical improvement measures at follow-up visits will include the ADHD-RS and the Clinical Global Impression- Improvement Scale (Guy, 1976). Once a change in the CGI-I score of < 2 or a decrease in the ADHD-RS score of 30% or greater is noted, we will not further increase the daily dosage.

Patients will return for 5 weekly visits. Vital signs, cardiac auscultation, and a routine follow-up physical examination will be performed at each visit.

Patients experiencing adverse effects that are judged by the investigator to be clinically significant, as well as non-serious but bothersome adverse effects that do not respond to dose adjustment will be taken off SRG. Events judged to be serious will be reported to the IRB, FDA, and Shire.

After 5 visits, subjects assessed as having had a significant improvement in the ADHD-RS or CGI-I will take the WJ-III "B" form (see above) beginning 2 hours after taking their current dose.

Data analysis:

The subjects' scores on the WJ-III, obtained initially and then during treatment with GXR, will be compared using a one-tailed t-test.

Continuation:

Patients who have benefited from the study drug will be given the option of continuing the medication, prescribed by the same physician, supplied commercially. If they elect not to continue, the study drug will be tapered off by 1 mg (daily dosage) per week.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of ADHD-inattentive or combined type.

Exclusion Criteria:

* Intelligence (IQ) below 85 as determined by formal testing.
* Identified or suspected genetic syndromes.
* Autism or other pervasive developmental disorders.
* Psychiatric disorders other than ADHD and oppositional defiant disorder.
* Heart, liver or renal disease.
* Cancer.
* Epilepsy or non-febrile seizure history.
* Cardiac arrhythmia, bradycardia, or syncope.
* Any other condition considered to be potentially exacerbated or endangered by treatment with an alpha-2 agonist drug.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
one-tailed t-test | 7 weeks
  Improvement in Woodcock Johnson III score when taking sustained release guanfacine, compared to score on the same test prior to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology Group of Bergen County, Ridgewood, New Jersey, United States

REFERENCES:
- [Background] 1. Shaywitz S, Beecher J, Shaywitz G. Issues in the definition and classification of attention deficit disorder. Topics in language disorders . 1994;14:1-25.. 2. Pastura G, Mattos P, Prufer A. Academic Performance in ADHD When Controlled for Comorbid Learning Disorders, Family Income, and Parental Education in Brazil. J J Att Dis. 2009;12:469-473 3. Barbaresi W, Katusic W, Slavica K et al. Modifier of long-term school outcomes for children with attention-deficit/hyperactivity disorder. Does treatment with stimulant medication make a difference? Results from a population based study.; J Devel Behav Pediatrics. 2007;28(4):274-287. 4. Forness S, Kavale K (2002): Impact of ADHD on School Systems. In: Jensen P and Cooper J, Attention Deficit Hyperactivity Disorder. Kingston NJ: Civic Research Inst.; 24-3 - 24-7. 5. Pliszka S, Carlson C, Wanson J (1999). Learning Disorders. In: ADHD with Comorbid Disorders. New York: Guilford Press; 188-201. 6. Gianarris W, Golden C, Greene L. The Conners' parent rating scales: a critical review of the literature. Clin Psychol Rev. 2001;21:1061-1093. 7. Scheffler RM, Brown TT, Fulton BD et al Positive association between attention deficit/hyperactivity disorder medication use and academic achievement during elementary school. Pediatrics 2009;123(5):1273-1279 8. Biederman J, Boellner S, Childress A et al. Lisdexamfetamine dimesylate and mixed amphetamine salts extended-release in children with ADHD: a double-blind, placebo-controlled, crossover analog classroom study. Biol Psychiatry 2007;62:970-976. 9. Pelham WE, Manos MJ, Ezzell CE, et al. A dose-ranging study of a methylphenidate transdermal system in children with ADHD. J Am Acad Child Adolesc Psychiatry 2005;44:522-9. 10. Mayes S, Calhous S. Frequency of reading, math, and writing disabilities in children with clinical disorders. Learning and Individual Differences. 2006;16:145-157.